CLINICAL TRIAL: NCT00007306
Title: Evaluation of the Therapeutic Efficacy & Safety of Topical Administration of Parathyroid Hormone (PTH) in Psoriasis
Brief Title: Treatment of Psoriasis With Parathyroid Hormone
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: R43AR046653 (NIH); NIAMS-059
Record Dates: First submitted 2000-12-16; First posted 2000-12-18 (Estimated); Last update posted 2007-01-04 (Estimated); Status verified 2003-03

CONDITIONS: Plaque Psoriasis
Keywords: Parathyroid hormone; Psoriasis; Lesions; Topical medications; Ointment; Calcium metabolism; Skin biopsy
MeSH Terms: conditions — Psoriasis

INTERVENTIONS:
Drug: Parathyroid hormone ointment

SUMMARY:
This is a clinical study in two phases. The first phase compares the effect of an ointment containing parathyroid hormone (PTH) with the effect of a placebo ointment (inactive ointment without PTH) on psoriasis lesions. Neither the study participants nor the researchers will know who is receiving PTH ointment and who is receiving placebo until the end of this first study phase. The second phase is a study of the PTH ointment on large areas of psoriasis to find out how long the effects last.

DETAILED DESCRIPTION:
Patients with active plaque psoriasis will be withdrawn from systemic and topical medications. After washout, we will select active psoriatic lesions of at least 25 square cm in size to receive either placebo ointment or a proprietary ointment containing PTH for 8 weeks. We will see the patients every 2 weeks. We will evaluate the lesions by examination and digital photography at each visit and measure parameters of calcium metabolism periodically during the 8 weeks.

At the conclusion of the 8 weeks, we will obtain punch biopsies from the treated lesions and from one lesion without treatment. If the patients elect, we will transition them into an open label trial with the PTH ointment including up to 1000 square cm of psoriatic lesions and monitor them for duration of effect and changes in parameters of calcium metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Active plaque psoriasis at least 10 percent BSA (body surface area)
* Age 18-70

Exclusion Criteria:

* Abnormalities of calcium metabolism

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2000-01; Study Completion 2005-04

CONTACTS AND LOCATIONS:
Overall Officials: Michael Holick, PhD, MD, Principal Investigator
Locations (1):
- Boston University School of Medicine, Boston, Massachusetts, United States

REFERENCES:
- [Background] Holick MF, Chimeh FN, Ray S. Topical PTH (1-34) is a novel, safe and effective treatment for psoriasis: a randomized self-controlled trial and an open trial. Br J Dermatol. 2003 Aug;149(2):370-6. doi: 10.1046/j.1365-2133.2003.05437.x. PMID 12932245